CLINICAL TRIAL: NCT03976258
Title: The Impact of Intravenous Heroin Use on Immune Activation in Treated HIV
Brief Title: Effect of Heroin Use on Immune Activation and Cardiovascular Risk in HIV
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Corrilynn Hileman, Principal Investigator, MetroHealth Medical Center
Other Study IDs: IRB17-00336 and IRB17-00429; 1R01DA044576-01 (NIH)
Record Dates: First submitted 2018-07-12; First posted 2019-06-05 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: HIV Infection; Opioid-use Disorder; Cardiovascular Diseases
Keywords: heroin; HIV; inflammation; cardiovascular
MeSH Terms: conditions — HIV Infections; Opioid-Related Disorders; Cardiovascular Diseases; Inflammation | interventions — Buprenorphine, Naloxone Drug Combination; Methadone; Naltrexone; vivitrol; Heroin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine, stool, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- HIV-infected adults actively using heroin: HIV-infected adults on antiretroviral therapy who are currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past.
  Interventions: Drug: Heroin
- HIV-infected adults never having used heroin: HIV-infected adults on antiretroviral therapy matched to HIV-infected adults actively using heroin by age, sex and CD4+ count.
- HIV-infected adults initiating buprenorphine/naloxone: HIV-infected adults on antiretroviral therapy who are currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past initiating medication assisted treatment (MAT) for opioid use disorder with buprenorphine/naloxone.
  Interventions: Drug: buprenorphine/naloxone
- HIV-uninfected adults initiating buprenorphine/naloxone: HIV-uninfected adults who are currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past initiating medication assisted treatment (MAT) for opioid use disorder with buprenorphine/naloxone.
  Interventions: Drug: buprenorphine/naloxone
- HIV-infected adults initiating methadone: HIV-infected adults on antiretroviral therapy who are currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past initiating medication assisted treatment (MAT) for opioid use disorder with methadone
  Interventions: Drug: Methadone
- HIV-infected adults initiating Vivitrol: HIV-infected adults on antiretroviral therapy who are currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past initiating medication assisted treatment (MAT) for opioid use disorder with Vivitrol.
  Interventions: Drug: Naltrexone Injection
- HIV-uninfected adults initiating methadone: HIV-uninfected adults who are currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past initiating medication assisted treatment (MAT) for opioid use disorder with methadone.
  Interventions: Drug: Methadone
- HIV-uninfected adults initiating Vivitrol: HIV-uninfected adults who are currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past initiating medication assisted treatment (MAT) for opioid use disorder with Vivitrol.
  Interventions: Drug: Naltrexone Injection

INTERVENTIONS:
Drug: buprenorphine/naloxone — This is an observational study. Buprenorphine/naloxone for opioid use disorder will be provided in a standardized way by experienced providers through already established funded treatment programs.
  Groups: HIV-infected adults initiating buprenorphine/naloxone; HIV-uninfected adults initiating buprenorphine/naloxone
Drug: Methadone — This is an observational study. Methadone for opioid use disorder will be provided in a standardized way by experienced providers through already established funded treatment programs.
  Groups: HIV-infected adults initiating methadone; HIV-uninfected adults initiating methadone
Drug: Naltrexone Injection — This is an observational study. Naltrexone injection for opioid use disorder will be provided in a standardized way by experienced providers through already established funded treatment programs.
  Other Names: Vivitrol
  Groups: HIV-infected adults initiating Vivitrol; HIV-uninfected adults initiating Vivitrol
Drug: Heroin — This is an observational study. Participants using heroin will be enrolled into this group.
  Groups: HIV-infected adults actively using heroin

SUMMARY:
Despite the advent of safer HIV therapies, high levels of markers of systemic inflammation and increased cardiovascular risk threaten the well-being of individuals living with HIV and present a significant challenge for HIV providers. These risks may be accentuated in HIV-infected individuals who are active intravenous drug users (IVDU); however, this population has been specifically excluded from prior studies assessing immune activation and cardiovascular risk in people living with HIV. In this study, the investigators will specifically target HIV-infected participants who are active IVDU, and co-enroll a control group of HIV-infected participants who never used IV drugs. The investigators will study the specific alterations in immune activation and several mechanisms felt to be potential drivers of immune activation outside of the IVDU population, namely gut integrity alteration, microbial translocation, and oxidized lipids. The investigators will also study the effect of IVDU on markers of arterial inflammation and vascular function. Importantly, the investigators will study the reversibility of immune activation, gut dysfunction, and cardiovascular markers after cessation of IVDU, and to that effect, compare strategies for IVDU cessation-buprenorphine/naloxone versus methadone or vivitrol maintenance treatment.

DETAILED DESCRIPTION:
This is a 48-week matched, prospective, observational, cohort study of HIV-infected adults on antiretroviral therapy who actively use heroin or who have never used heroin. The overarching goals are 1) to define the extent and specifics of immune activation in HIV-infected IV heroin users; 2) to define the effect of IV heroin on gut integrity and permeability, and the relationship of gut integrity alteration and immune activation; 3) importantly, to study the reversibility of immune activation, inflammation, and gut dysfunction after cessation of IV heroin, and to that effect, compare strategies for medication assisted treatment-buprenorphine/naloxone versus methadone or vivitrol maintenance; 4) to study if heightened immune activation associated with active intravenous drug use (IVDU) is associated with higher cardiovascular disease risk, including endothelial dysfunction and arterial inflammation, and if these effects are reversible with buprenorphine/naloxone or methadone.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection or no HIV infection
* 18 years or older
* HIV-1 RNA < 400 if HIV-infected and on antiretroviral therapy
* On stable antiretroviral therapy at least 12 weeks with cumulative duration of at least a year for HIV-infected if on antiretroviral therapy
* Currently using heroin at least 1 month with a cumulative duration of at least 12 months in the past for active heroin group
* Initiating medication assisted treatment for active heroin use initiating medication assisted treatment groups

Exclusion Criteria:

* Active infection, malignancy or other inflammatory condition
* Uncontrolled diabetes or hypothyroidism
* Known cardiovascular disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adults ages 18 to 80 years with and without HIV infection using heroin or initiating treatment for heroin use or not using heroin.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in plasma soluble CD14 concentration | 48 weeks
  soluble marker of monocyte activation
Change in Endopat measure of microvascular function | 48 weeks
  Measure of endothelial function
Change in target to background ratio measured by fluorodeoxyglucose (FDG)-positron emission tomography (PET) | 48 weeks
  Measure of vascular inflammation
Change in plasma Interferon Gamma-Induced Protein 10 concentration | 48 weeks
  soluble marker of inflammation
Change in plasma intestinal fatty acid binding protein concentration | 48 weeks
  soluble marker of gut integrity

SECONDARY OUTCOMES:
Change in total fat stores measured by Whole body Dual-energy X-ray absorptiometry | 48 weeks
  Measurement of fat stores
Change in aortofemoral pulse wave velocity | 48 weeks
  Measure of arterial stiffness
Change is waist to hip ratio | 48 weeks
  Measurement of central obesity
Change in body mass index | 48 weeks
  Body measurement

CONTACTS AND LOCATIONS:
Overall Officials: Corrilynn O Hileman, MD, Principal Investigator — MetroHealth Medical Center; Grace A McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Metrohealth Medical center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No